CLINICAL TRIAL: NCT01527877
Title: An Open Label, Single Arm, Multicenter Phase II Study of BKM120 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck Who Failed to Respond to Platinum-based Therapy
Brief Title: Study of BKM120 in Advanced Squamous Cell Carcinoma of Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Byoung Chul Cho, Assistant professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0828-001
Record Dates: First submitted 2012-01-26; First posted 2012-02-07 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Head Neck Cancer Squamous Cell Metastatic; Head Neck Cancer Squamous Cell Recurrent
Keywords: BKM120; head and neck cancer; squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — Patients will be instructed to take BKM120 orally at a dose of 100 mg with a glass of water once daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day. The patient will be dosed on a flat scale of mg/day and not be adjusted to body weight or body surface area. If vomiting occurs no attempt should be made to replace the dose.
  • BKM120 should be taken 1-hour following a light meal. Please note that patients must avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction. Regular orange juice is allowed.
  Other Names: NVP-BKM120; BKM-120

SUMMARY:
This study is to evaluate disease control rate (DCR) at 8 weeks of BKM120 administered as therapy for patient with recurrent/metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
One promising approach to the treatment of cancer is inhibition or modulating the crucial signal transduction pathway of PI3K-Akt-mTOR. Several PI3K inhibitors are being tested in the clinical trials for cancer treatment but not for the head and neck cancer yet. BKM120 is a specific Pan-class I PI3K inhibitor. We suggest multicenter single arm phase II study to determine anti-tumor effects of BKM120 in patients with recurrent and/or metastatic SCCHN who failed to prior platinum-based chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic squamous-cell carcinoma of head and neck (SCCHN), except nasopharyngeal carcinoma
* Disease not amenable to curative treatment (surgery or radiation for curative intent)
* 20 years of age or older
* Progressive disease defined as follows

  * after one or two prior chemotherapy regimens including platinum-based chemotherapy given for palliation
  * within 6 months after concurrent chemoradiotherapy (including induction chemotherapy) delivered as part of primary treatment.
* Life expectancy of at least 12 weeks
* At least one measurable lesion according to the RECIST 1.1 criteria.
* ECOG performance score of 0 ~ 2
* Adequate organ function

  * Absolutely Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hemoglobin ≥ 9.0 g/dL
  * Serum Creatinine ≤ 1.5 x ULN
  * Adequate liver function (total bilirubin ≤ 2.0 x ULN, AST and ALT ≤ 2.0 x ULN or < 5.0 x ULN if liver metastases are present)
* Availability of tissue samples (archival tissue or rebiopsied tissues) for molecular analysis (representative paraffin block or unstained sections from tumor diagnostic specimen are mandatory)
* Patients who have will and ability to comply with the scheduled visits, the treatment plan, laboratory tests and any other trial procedures
* Patient's informed consent

Exclusion Criteria:

* Nasopharyngeal carcinoma
* More than two prior lines of chemotherapy in the palliative setting.
* Uncontrolled, untreated brain metastasis Patients with controlled and asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases ≥ 28 days (must include radiotherapy and/or surgery) and, if on corticosteroid therapy, should be receiving a stable low dose (e.g. dexamethasone 4 mg or equivalent dose of another corticosteroid for at least 14 days before start of study treatment)
* Surgery, chemotherapy or irradiation within 4 weeks of study entry
* Prior treatment with any investigational drug within the preceding 4 weeks
* Concomitant chemotherapy, hormonal therapy or immunotherapy
* Previous or concomitant malignant disease, except adequately treated basal cell cancer of the skin or cervical cancer in situ, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 5 years prior study entry
* Patient who cannot take the oral drug
* Patient is pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Clinically significant psychological disorders including mood and anxiety disorders judged by psychiatry physician
* Patient who have not recovered to grade 1 or better from any adverse events (except alopecia) related to previous antineoplastic therapy before screening procedures are initiated
* Severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

  * Patient has poorly controlled diabetes mellitus (HbA1c> 8 %)
  * Patient has history of cardiac dysfunction including history of documented congestive heart failure (New York Heart Association functional classification III-IV) and documented cardiomyopathy
  * Patient is currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes. * Active infection, inflammatory bowel disease
  * Inadequate liver function (total bilirubin ≥ 2.0 x ULN, AST and ALT ≥ 2.0 x ULN or ≥ 5.0 x ULN if liver metastases are present)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Disease control rate at 8 weeks | Eight weeks after administration of the drug
  The disease control rate (DCR) is defined as the proportion of randomized patients achieving a best overall response of PR or CR or SD, defined by RECIST criteria (version 1.1), relative to the total number of patients in the considered analysis population (ITT).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Every 8 weeks from date of first treatment until date of last treatment up to 24 months
  Overall objective response rate (ORR) is the best response rate stipulated as complete response (CR) or partial response (PR) (target lesion and tumor response defined according to RECIST guideline version 1.1) and identified as percentage of the confirmed patients.
Toxicity profile | Every 4 weeks from date of first treatment until date of last treatment up to 24 months
  From C1D1 to 1 months after the last dose adminitration
  Overall safety profile verified as relevance of adverse events and laboratory abnormality in the study and grades granted based on (USA National Cancer Center) Common Terminology Criteria for Adverse Events such as the type, frequency and severity (CTCAE), v4.0.
Overall survival | Every 8 weeks from date of first treatment until the date of death from any cause, assessed approximately up to 24 months
  From C1D1 to death
Progression-free survival | Every 8 weeks from date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 24 months
  From C1D1 until confirmed disease progression or death
Quality of life assessment | Every 4 weeks from date of first treatment until the date of death from any cause, assessed approximately up to 24 months
  Quality of life assessment will be performed using FACT-HN& questionnaire
  FACT-H&N questionnaire includes physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and head & neck cancer subscale (HNCS).
  Patients will be evaluation on baseline, day 1 of every cycle (4 weeks), and end of treatment.
Time to progression (TTP) | Every 8 weeks from date of first treatment until the date of first documented progression, assessed approximately up to 24 months
  From C1D1 until confirmed disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Chul Cho, M.D., Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HR, Kang HN, Yun MR, Ju KY, Choi JW, Jung DM, Pyo KH, Hong MH, Ahn MJ, Sun JM, Kim HS, Kim J, Yoo J, Kim KR, Koh YW, Kim SH, Choi EC, Yoon SO, Shim HS, Paik S, Kim TM, Cho BC. Mouse-human co-clinical trials demonstrate superior anti-tumour effects of buparlisib (BKM120) and cetuximab combination in squamous cell carcinoma of head and neck. Br J Cancer. 2020 Dec;123(12):1720-1729. doi: 10.1038/s41416-020-01074-2. Epub 2020 Sep 23. PMID 32963347